CLINICAL TRIAL: NCT05991622
Title: Integrating Long-Acting Injectable Treatment to Improve Medication Adherence Among Persons Living With HIV and Opioid Use Disorder
Brief Title: Combined Injectable Treatment for HIV and OUD
Acronym: CHOICE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Josiah Rich, Principal Investigator, Rhode Island Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA055498 (NIH)
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Human Immunodeficiency Virus; Opioid Use Disorder
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Opioid-Related Disorders | interventions — Sublocade; Rilpivirine; cabotegravir, rilpivirine drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Preliminary Test of Combined LAI Treatment (Experimental): The combined injectable treatment includes a dual-administration of rilpivirine (CAB/RPV) "cabenuva" for HIV and extended-release buprenorphine (XR-B) "sublocade" for OUD.
  Interventions: Drug: Combined LAI Treatment: Cabenuva and Sublocade

INTERVENTIONS:
Drug: Combined LAI Treatment: Cabenuva and Sublocade — A preliminary test of the combined LAI treatment will be conducted with a total of 30 individuals diagnosed with HIV and OUD that meet all other study inclusion criteria. Treatment will take place primarily at TMH IC (n=30). Participants deemed fit for the study (per recommendation by TMH IC staff and subsequent medical chart review) will receive the combined LAI treatment (described below), and complete follow-up assessments at 1-, 3-, and 6-months following initiation of injectable medication. Of the 30 participants, 25 will be purposefully selected to engage in qualitative interviews to assess the strengths and limitations of the clinical protocol and combined treatment as well as describe their reasons for LAI uptake or discontinuation. We will also elicit feedback from clinic staff and other key stakeholders regarding the delivery of the clinical protocol and other implementation factors
  Other Names: rilpivirine (CAB/RPV) "cabenuva"; extended-release buprenorphine (XR-B) "sublocade"

SUMMARY:
This is study seeks to evaluate perspectives of a combined injectable treatment for HIV and OUD. Specifically, with the development of new long-acting medications such as cabotegravir co-administered with rilpivirine (CAB/RPV) and extended-release buprenorphine (XR-B) there is a need to better understand factors that influence the delivery and uptake of this type of treatment. The current study seeks to conduct a single-arm open pilot trial of a clinical protocol and implementation approach for the combined HIV/OUD LAI treatment. Participants will include patients receiving treatment at TMH IC (n=30) and clinic staff (n=5-10). Participants will complete a baseline survey, receive the combined LAI treatment, and complete follow-up assessments at 1-, 3-, and 6-months following initiation of injectable medication. Of the 40 participants, 25 will be purposefully selected to engage in qualitative interviews to assess the strengths and limitations of the clinical protocol and combined treatment as well as describe their reasons for LAI uptake or discontinuation.

DETAILED DESCRIPTION:
Treatment services for HIV and OUD have historically been delivered across multiple settings leading to fragmented and uncoordinated care. Models of behavior change suggest that addressing multiple health conditions simultaneously through integrated, evidence-based, interventions has the potential to overcome traditional barriers to optimize engagement and improve clinical outcomes. Consistent with this perspective, numerous studies have documented that receipt of opioid agonist treatment, in the context of HIV care, is associated with ART adherence and decreased HIV viral loads. Recent pharmacological advancements have led to the development of novel long-acting, injectable, medications for HIV [cabotegravir co-administered with rilpivirine (CAB/RPV)] and OUD (extended-release buprenorphine). These therapies have the potential to dramatically improve adherence, lead to better control of both diseases, and reduce mortality rates for this vulnerable population. However, currently, little is known about 1) the perceived acceptability/feasibility of combining HIV and OUD treatment into a single point of care; and 2) how best to deliver integrated, monthly injectable, treatment for HIV and OUD to facilitate future implementation. The long-term goal of this line of research is to disseminate an efficacious, integrated, injectable treatment program for HIV and OUD. Through formative qualitative evaluation, our team developed the clinical protocol and implementation procedures for the combine HIV and OUD care using long-acting injectable therapies. As such, the present study is recruiting TMH IC patients (n=30) and clinical staff (n=5-10) for a single-arm open pilot trial of the clinical protocol to determine the effectiveness of implementation strategies for the combined LAI treatment. The investigators expect that, as a result of this project, the protocol will demonstrate high degrees of feasibility, acceptability, and uptake of long-acting injectable medications for HIV and OUD. This work will serve as the foundation for a future NIH Hybrid Type 1 Effectiveness-Implementation study.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay
* Current diagnosis of OUD according to DSM-5
* Able to understand and speak English and to provide written and verbal informed consent

Exclusion Criteria:

* Currently pregnant, breastfeeding, planning to become pregnant or breastfeed during the study period
* Coinfection of Hepatitis B or plans to get treated for Hepatitis C during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | 6 months
  percent of patients interested in the treatment, patient eligibility rate, consent rate, rate of recruitment, percent of participants who initiate injectables, follow-up completion rate (through 6 months), and reasons for refusal
Acceptability | 6 months
  study dropout rate (those who were lost to follow-up) and rate of discontinuation of injectables (those who decided to transition back to oral/sublingual regimen) as indices of
Feasibility/Acceptability | 6 months
  Client Satisfaction Questionnaire-Revised: assess consumer satisfaction with health and human services including governmental and public benefit programs and services
Self-report of engagement in treatment | 6 months
  Treatment Effectiveness Assessment : elicits patient responses that help the patient and the clinician quickly gauge patient progress in treatment and in recovery, according to the patients' sense of what is important within four domains -- substance use, health, lifestyle, community,
Feasibility/Acceptability | 6 months
  Qualitative interviews to explore the acceptability and feasibility of the intervention format (e.g. processes and procedures, access to support services, tolerability of medication) and how the intervention could be strengthened, identifying areas needing refinement or improvement for future iterations.

SECONDARY OUTCOMES:
Substance use | 6 months
  National Epidemiologic Survey on Alcohol and Related Conditions (NESARC)
Substance use | 6 months
  NIDA-modified ASSIST - tool to identify risky substance use
Substance use | 6 months
  urine drug screens from the individual's electronic medical record
HIV Risk Behavior | 6 months
  Texas Christian University (TCU) HIV/AIDS Risk Assessment: a measure of overall sex and drug risk behavior
Treatment services | 6 months
  Treatment Services Review will be used to assess receipt of case management, psychiatric, peer recovery coaching, and other treatment services, including utilization of other medications for OUD (e.g., if a participant has transitioned to Methadone).
Overall Quality of life | 6 months
  Q-LES-Q-SF, a psychometrically sound shorter version of the original Q-LES-Q. It consists of a self-reported 16-item questionnaire that has shown internal consistency, rest-retest reliability, and convergent and criterion validity (80% sensitivity, 100% specificity)

CONTACTS AND LOCATIONS:
Overall Officials: Josiah D Rich, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT05991622/ICF_000.pdf